CLINICAL TRIAL: NCT01867905
Title: The Effect of Antibiotic Administration on Blood Culture Positivity in Patients With Severe Sepsis and Septic Shock: a Prospective Multicenter Observational Trial.
Brief Title: Antibiotic Administration and Blood Culture Positivity in Severe Sepsis and Septic Shock
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: McGill University (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Matthew Pellan Cheng, Medical Resident, University of British Columbia
Other Study IDs: H12-01716; H12-01716
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Severe Sepsis; Septic Shock; Bacteremia
Keywords: Severe sepsis; Septic shock; Bacteremia; Antibiotics; Blood culture positivity
MeSH Terms: conditions — Sepsis; Shock, Septic; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cultures
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe sepsis and septic shock: Patients who present in severe sepsis or septic shock will have blood cultures taken before and after antibiotic administration. The antibiotic choice will be determined by the emergency physician and the patients will be treated as per routine hospital protocol. No therapeutic interventions will be administered.

SUMMARY:
Sepsis is a significant cause health care expenditure and carries an extremely high rate of morbidity and mortality if not treated appropriately. From 1979 to 2000, sepsis resulted in over 10 million admissions to hospital in the United States with a mortality rate of 17.9 to 27.8 percent. In Canada, it is estimated that the incidence of sepsis from 2008-2009 was 103.3 per 100,000 per year.

Advances in the multifaceted management of sepsis in recent years have resulted in improved clinical outcomes. However, the cornerstone of sepsis management relies on the prompt administration of appropriate antibiotics. Current clinical practice suggests that antibiotic administration can be delayed up to 45 minutes in order to obtain blood cultures, whose results have a profound impact on the type and duration of antimicrobial therapy. Unfortunately, this recommendation is based on very little evidence and the investigators have found that potential life-saving treatment is often delayed in order to abide by it. Furthermore, recent data suggest that mortality could be increased by approximately 5% by delaying antibiotic administration for that time period.

The investigators therefore wish to organize a prospective, multi-centre trial in order to identify the effect of antibiotic administration on blood culture positivity in patients presenting with severe sepsis or septic shock. Other objectives will be to elucidate which patient factors, including age, co-morbid conditions and clinical presentation, as well as antibiotic choice will affect blood culture results.

This study will be conducted in the emergency departments at St. Paul's Hospital (SPH), Vancouver General Hospital (VGH), Lion's Gate Hospital (LGH), Surrey Memorial Hospital, Montreal General Hospital (MGH), Royal Victoria Hospital (RVH) and Maricopa Integrated Health System. Patients identified for the aforementioned conditions will be treated as per routine hospital protocol. If the patient is deemed eligible for the study, a second set of blood of blood cultures will subsequently be drawn ideally between 30 and 60 minutes after the administration of antibiotic therapy. Subject demographic data will be collected pertaining to age, comorbid immunocompromised conditions, vital signs, laboratory tests pertaining to end organ dysfunction, suspected source of sepsis, the type antibiotics administered and the timing of antimicrobial administration with respect to the second set of blood cultures taken.

Our hypothesis is that blood culture positivity in patients presenting with severe sepsis and septic shock will not be altered significantly by antibiotic therapy. If so, our study would strongly argue against delaying life-saving therapy and would thus greatly improve patient care in our local emergency rooms. If incorrect, our study would be the first to demonstrate the benefit of obtaining blood cultures before antibiotic therapy and would strengthen current recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age who present to the emergency department with the diagnosis of severe sepsis/septic shock.
* This will include patients that have 2/4 systemic inflammatory response syndrome criteria, a suspected infection and either a initial serum lactate > 4mmol/L or a initial systolic blood pressure < 90 millimeters of mercury.

Exclusion Criteria:

* Patients in whom antibiotics have been administered >2 hours prior to assessment.
* Patients with antibiotics in the community in the past 48 hours
* Patients with known severe coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age > 18) who present to the emergency department with severe sepsis/septic shock .
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
The effect of antibiotic administration on blood culture positivity in patients with severe sepsis and septic shock: a prospective multicenter observational trial. | Four months
  The primary outcome is the measure of blood culture positivity before and after antibiotic administration.

CONTACTS AND LOCATIONS:
Overall Officials: David Sweet, M.D., Principal Investigator — University of British Columbia
Locations (7):
- Maricopa Integrated Health Center, Phoenix, Arizona, United States
- Canada (6):
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Saint-Paul's Hospital, Vancouver, British Columbia
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Paquette K, Sweet D, Stenstrom R, Stabler SN, Lawandi A, Akhter M, Davidson AC, Gavric M, Jinah R, Saeed Z, Demir K, Sangsari S, Huang K, Mahpour A, Shamatutu C, Caya C, Troquet JM, Clark G, Wong T, Yansouni CP, Cheng MP. Neither Blood Culture Positivity nor Time to Positivity Is Associated With Mortality Among Patients Presenting With Severe Manifestations of Sepsis: The FABLED Cohort Study. Open Forum Infect Dis. 2021 Jun 17;8(7):ofab321. doi: 10.1093/ofid/ofab321. eCollection 2021 Jul. PMID 34307728
- [Derived] Cheng MP, Stenstrom R, Paquette K, Stabler SN, Akhter M, Davidson AC, Gavric M, Lawandi A, Jinah R, Saeed Z, Demir K, Huang K, Mahpour A, Shamatutu C, Caya C, Troquet JM, Clark G, Yansouni CP, Sweet D; FABLED Investigators. Blood Culture Results Before and After Antimicrobial Administration in Patients With Severe Manifestations of Sepsis: A Diagnostic Study. Ann Intern Med. 2019 Oct 15;171(8):547-554. doi: 10.7326/M19-1696. Epub 2019 Sep 17. PMID 31525774